CLINICAL TRIAL: NCT01264146
Title: Hyperbaric Oxygen Therapy in Calcaneal Intraarticular Fractures: Can it Decrease the Soft-tissue Complication Rate?
Acronym: HOCIF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTC-A10-025
Record Dates: First submitted 2010-12-17; First posted 2010-12-21 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Microcirculation; Wound Healing
Keywords: hyperbaric oxygen therapy; calcaneal fracture; calcaneal plating; wound infection; microcirculation
MeSH Terms: conditions — Wound Infection | interventions — Hyperbaric Oxygenation; salicylhydroxamic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- calcaneal plating HBOT (Active Comparator): Open reduction and internal fixation of calcaneal fracture + HBOT
  Interventions: Procedure: HBOT
- calcaneal plating (Placebo Comparator): Open reduction and internal fixation of calcaneal fracture + Placebo (Sham)
  Interventions: Procedure: Placebo (Sham)

INTERVENTIONS:
Procedure: HBOT — Open reduction and internal fixation of calcaneal fracture + hyperbaric oxygen therapy 20 postoperative days (one time, 90 minutes a day)
  Other Names: calcaneal plating; hyperbaric oxygen therapy
  Arms: calcaneal plating HBOT
Procedure: Placebo (Sham) — open reduction and internal fixation of calcaneal fracture + Placebo (Sham)
  Other Names: calcaneal plating; Sham procedure (HBOT)
  Arms: calcaneal plating

SUMMARY:
This study aims to test the hypothesis that postoperative daily hyperbaric oxygen therapy (HBOT) decreases soft-tissue complication rate during the operative handling of intra-articular calcaneal fractures. Minor motivations: 1. To evaluate microcirculatory criteria of cutaneous tissue predicting emerging wound healing defects, 2. To identify patients at risk for soft-tissue complication after calcaneal plate osteosynthesis and to determine the optimal time point for operative intervention using these microcirculatory criteria preoperatively, 3. To evaluate the effect of HBOT on postoperative microcirculation, 4. To collect preliminary data to evaluate the economical impact of wound complications, with and without HBOT, 5. To identify a correlation between HBOT with expected limited soft-tissue complication rate and the clinical and radiographic outcome two years after surgery.

DETAILED DESCRIPTION:
Wound complication remains an important problem in calcaneal fractures, with some plate series quoting up to a 27% infection rate. The original hypothesis stimulating this study is that HBOT after calcaneal plating can decrease such high rates of infection. Validation of this hypothesis would not only alter guidelines for standard procedure (plate osteosynthesis), but would also help to avoid difficult follow-up operations and improve functional outcome after calcaneal fracture. To date, this therapeutic approach has not been systematically tested in the existing literature. As further motivation for this study, the assessment of the existent microcirculation as a potential screening parameter will be analysed. In order to do so, it is assumed that wound infection partially develops due to disruptions in the microcirculation. This leads to the hypotheses, that by measuring the microcirculation, patients at high risk for post operative infections could be identified before operation, planning a different less invasive approach or conservative treatment.

ELIGIBILITY:
Inclusion Criteria:

* Acute displaced intraarticular calcaneal fracture

Exclusion Criteria:

* Extraarticular or open fracture, re-fracture or past surgical procedures in calcaneal region, peripheral vascular disease, insulin dependent diabetes mellitus, macroangiopathy: Study population is representative for all calcaneal fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Postoperative rate of wound complication after calcaneal plating | 30 days
  Rate of postoperative wound edge necrosis and superficial or deep infection determined by wound redness, secretion of pus, detection of a microbial agens, CRP elevation and detection of fluid by sonography.

SECONDARY OUTCOMES:
Effect of HBOT on postoperative microcirculation of the foot, clinical outcome | 2 years
  Complications later than day 20 post-surgery, clinical and radiographic outcome (2years follow-up), To evaluate microcirculatory criteria of cutaneous tissue, To identify patients at risk for soft-tissue complication after calcaneal plate osteosynthesis and to determine the optimal time point for operative intervention, To evaluate the effect of HBOT on postoperative microcirculation, To identify a correlation between HBOT with expected limited soft-tissue complication rate and the clinical and radiographic outcome two years after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Knobe, MD, Principal Investigator — Dpt. of Orthopedic Trauma, RWTH Aachen University; Hans-Christoph Pape, MD, Study Chair — Dpt. of Orthopedic Trauma, RWTH Aachen University
Locations (1):
- RWTH Aachen University, Aachen, Germany

REFERENCES:
- [Derived] Lichte P, Blasius FM, Ganse B, Gueorguiev B, Pastor T, Nebelung S, Migliorini F, Klos K, Modabber A, Scaglioni MF, Schopper C, Hildebrand F, Knobe M. Intraoperative pneumatic tourniquet application reduces soft-tissue microcirculation, but without affecting wound healing in calcaneal fractures. Eur J Med Res. 2024 Sep 17;29(1):462. doi: 10.1186/s40001-024-01996-0. PMID 39289760
- [Derived] Knobe M, Iselin LD, van de Wall BJM, Lichte P, Hildebrand F, Beeres FJP, Link BC, Gueorguiev B, Nebelung S, Ganse B, Migliorini F, Klos K, Babst R, Haefeli PC. Reduced pre-operative skin oxygen saturation predicts revision after open reduction and internal fixation in calcaneal fractures : A reduced pre-operative oxygen saturation as measured by laser-Doppler spectrophotometry in 8 mm depth is associated with revision surgery after open reduction and internal fixation of calcaneal fractures through an extended lateral approach. Int Orthop. 2021 Sep;45(9):2355-2363. doi: 10.1007/s00264-021-05157-4. Epub 2021 Aug 6. PMID 34357432